CLINICAL TRIAL: NCT02464020
Title: A Pilot Study to Characterize Bile Acid Metabolism and Dysbiosis in Primary Sclerosing Cholangitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GI-2015-23049
Record Dates: First submitted 2015-05-29; First posted 2015-06-08 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Primary Sclerosing Cholangitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Cholangitis, Sclerosing; Inflammatory Bowel Diseases | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primary sclerosing cholangitis (Experimental): Two week course of oral vancomycin 500mg twice a day.
  Interventions: Drug: Vancomycin
- Control group (No Intervention): A control group of participants without Primary Sclerosing Cholangitis. Control group will consist of both healthy subjects and subjects with Inflammatory Bowel Disease.

INTERVENTIONS:
Drug: Vancomycin — Oral vancomycin: 500mg suspended in prefilled syringes for oral use
  Arms: primary sclerosing cholangitis

SUMMARY:
The goal of this study is to assess if oral vancomycin can restore the normal bile acid metabolism of people with Primary Sclerosing Cholangitis and Inflammatory Bowel Disease. Study participants will provide blood and stool samples in order to evaluate the bile acid metabolism before a short course of vancomycin and then again after to assess for change. The investigators will also assess the blood and stool of healthy people, and people with IBD (without PSC) as a control group.

DETAILED DESCRIPTION:
Primary Sclerosing Cholangitis (PSC) is a chronic inflammatory and fibrotic disease of the intra and extrahepatic ducts of unknown etiology that predominately occurs in people with Inflammatory Bowel Disease (IBD). One hypothesis is that altered microbiome (bacteria in the gut) in people with IBD are responsible for the inflammation in the liver seen in PSC. Bile acids (BAs) represent a unique mechanism of communication between the host and intestinal microbiome and the liver. Synthesized in the liver, bile acids are metabolized by intestinal bacteria hydroxylases to secondary BAs which then re-enter the portal circulation. Altered metabolism of BAs has been associated with gallstones and colorectal cancer and is hypothesized to play a role in the inflammatory response of certain disease such as IBD and PSC.

IBD has been associated with impairment of bile acid (BA) metabolism. In addition BAs play a role in regulating bacterial growth of the intestine and thus have an effect on the integrity of the intestinal mucosa, which is an essential component of IBD. Perturbations in this system could increase bacterial translocation into the portal system due to loss of protective mucosal factors or bacterial overgrowth.

The overall goal of this study is to assess the changes in BAs metabolism following administration of oral vancomycin. The investigators will also describe the relationship of the intestinal microbiome and BA metabolism in PSC/IBD.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of PSC made by typical clinical, radiographic and biochemical criteria.
* Diagnosis of PSC > 3 months

Exclusion Criteria:

* Antibiotic use within 30 days of initial study visit
* Probiotic use within 30 days of initial study visit
* Extensive ileal disease
* Severe of fulminant IBD
* Diabetes and/or metabolic syndrome
* Chronic disease state deemed unacceptable for the study per investigator review
* Decompensated Cirrhosis
* Females who are pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Fecal bile acid composition | 5 days
  Fecal samples will be collected over 1 week. Bile acids will be measured on each sample and the average composition of primary to secondary bile acids over the 5 day period will be assessed. Comparison will be made pre and post vancomycin

SECONDARY OUTCOMES:
Microbiome diversity analysis | 5 days
  Fecal samples collected over the course of a week will be assessed by 16S r-Ribosomal Ribonucleic Acid gene profiling. Intestinal microbial communities will be assessed pre and post vancomycin administration.

CONTACTS AND LOCATIONS:
Overall Officials: Byron P Vaughn, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States